CLINICAL TRIAL: NCT03580252
Title: Reliability of Hammersmith Examination in Prediction of Neurological Outcomes In Preterm Infants - Observational Study (REHAPENO)
Brief Title: Reliability of Hammersmith Examination in Prediction of Neurological Outcomes (REHAPENO)
Acronym: REHAPENO
Status: Completed | Type: Observational
Sponsor: Abha International Private Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Fleifel001
Record Dates: First submitted 2018-04-19; First posted 2018-07-09 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Child Development Disorders; Preterm Infant; Cerebral Palsy
Keywords: preterm; Child Development Disorders; Hammersmith; neurological outcomes; epidemiology
MeSH Terms: conditions — Developmental Disabilities; Premature Birth; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm Infant Neurological Follow-Up: Preterm infants <37 weeks' gestational age (GA) at birth admitted to the neonatal nurseries at the Abha Private Hospital in Kingdom of Saudi Arabia. This project aims to recruit 50 infants <37weeks at birth over a 1-year stating from march 2018.
  A Correlation analyses for the outcomes with initial regular medical practice of MRI/Ultrasound and Hammersmith assessment.
  Interventions: Other: Correlation analyses for the outcomes

INTERVENTIONS:
Other: Correlation analyses for the outcomes — No medical intervention would be done. The single arm would receive regular practice of Hammersmith Assessment and MRI / Ultrasound

SUMMARY:
In this study workers are trying to test the correlation between Hammersmith Infant Neurological Examination and MRI brain/cranial ultrasound with early prediction of neurological developmental outcome of preterm neonates. This study is prospective cross-sectional collecting the data of patients according to daily standard medical practice

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate the neurobehavioural performance of infants born preterm using the Hammersmith Infant Neurological Examination (HINE) in standard medical practice and compare it with the gold standard MRI and ultrasound imagings. It would be possible to check do we need to use all the 3 examinations or Hammersmith examination would be enough reliable predictor. Secondary aim is to explore the relationships between MRI brain /cranial us abnormalities and HINE at term-equivalent age in infants born preterm in prediction of neurological outcome at 1 year of chronological age.

This study will be only single arm/single group. This group would receive the regular practice of MRI, Ultrasound (US) and Hammersmith assessments. The 3 assessments would be compared in relationships with the neonatal developmental outcomes (developmental milestones).

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants <37 weeks' GA at birth admitted to the neonatal nurseries at the Abha Private Hospital in Kingdom of Saudi Arabia. This project aims to recruit 50 infants <37weeks at birth over a 1-year stating from march 2018

Exclusion Criteria:

* -infants with congenital or chromosomal abnormalities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preterm infants <37 weeks' GA at birth admitted to the neonatal nurseries at the Abha Private Hospital in Kingdom of Saudi Arabia. This project aims to recruit 50 infants <37weeks at birth over a 1-year stating from march 2018
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Non inferiority of MRI to Hammersmith assessments in developmental outcomes | 12 month
  Hammersmith assessment will be tested for non-inferiority to gold standard assessment method by MRI in terms of sensitivity for early prediction of delayed neurological syndrome (DNS)

SECONDARY OUTCOMES:
Superiority testing for Hammersmith assessment to gold standard MRI | 12 month
  Testing the superiority of Hammersmith assessment versus gold standard MRI in terms sensitivity for early prediction of DNS
Comparing the correlations of MRI and US scans with early prediction of DNS | 12 month
  Comparing the correlations of MRI and US scans with the early prediction of DNS
Comparing the correlations of US scan and Hammersmith assessment | 12 month
  Comparing the correlations of US scan and Hammersmith assessment with the early prediction of DNS
Hammersmith health economic analyses if primary endpoint is achieved | 12 month
  Both cost minimization analyses and cost effective analyses would be applied
Specificity and sensitivity for all techniques MRI, US and Hammersmith | 12 month
  Calculations for specificity and sensitivity would be applied for MRI, US and Hammersmith

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Fleifel, MD MSc PhD, Study Chair — College of Medicine, Mansoura University; Rawya Abdelghani, MD MSc PhD, Study Director — College of Medicine, Al Azhar University; Mohamed Ameen, MICR RPh, Principal Investigator — IQVIA Switzerland
Locations (1):
- Abha Private Hospital, Abhā, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided